CLINICAL TRIAL: NCT03749577
Title: Nutritional Strategies to Increase Nitric Oxide Signaling in Raynaud's Phenomenon
Acronym: NivOSe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC17.270
Record Dates: First submitted 2018-07-03; First posted 2018-11-21 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Raynaud Phenomenon
Keywords: l-citrullin; beetroot juice; Raynaud's phenomenon
MeSH Terms: conditions — Raynaud Disease | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- L-citrulline (Experimental): Six cycles will be conducted over two consecutive winters. One cycle will consist of two 2-week supplementation periods.
  A 7 days wash-out period will be imposed between treatment periods (placebo and treatment).
  Interventions: Dietary Supplement: L-citrulline
- Beetroot juice (Experimental): Six cycles will be conducted over two consecutive winters. One cycle will consist of two 2-week supplementation periods.
  A 7 days wash-out period will be imposed between treatment periods (placebo and treatment).
  Interventions: Dietary Supplement: Beetroot juice
- L-citrulline placebo (Placebo Comparator): Six cycles will be conducted over two consecutive winters. One cycle will consist of two 2-week supplementation periods.
  A 7 days wash-out period will be imposed between treatment periods (placebo and treatment).
  Interventions: Dietary Supplement: L-citrulline placebo
- Denitrated beetroot juice (Placebo Comparator): Six cycles will be conducted over two consecutive winters. One cycle will consist of two 2-week supplementation periods.
  A 7 days wash-out period will be imposed between treatment periods (placebo and treatment).
  Interventions: Dietary Supplement: Denitrated beetroot juice

INTERVENTIONS:
Dietary Supplement: L-citrulline — L-citrulline 9g per day (capsule, per os) during 14 days;
  Arms: L-citrulline
Dietary Supplement: Beetroot juice — Concentrated 70 ml beetroot juice bottles containing 6.45 mmol of nitrates
  Arms: Beetroot juice
Dietary Supplement: L-citrulline placebo — L-citrulline placebo (maltodextrin) 9g per day (capsule, per os) during 14 days
  Arms: L-citrulline placebo
Dietary Supplement: Denitrated beetroot juice — Concentrated 70 ml nitrate-depleted beetroot juice
  Arms: Denitrated beetroot juice

SUMMARY:
The investigators aim at comparing the efficacy of a 2 weeks supplementation by L-citrulline or beetroot juice to L-citrulline placebo or denitrated beetroot juice respectively on Raynaud's phenomenon severity. Raynaud's phenomenon severity will be assessed through the Raynaud Condition Score, daily frequency of attacks or cumulative attack duration (expressed as min) daily collected by patients in a diary. Each Volunteer will choose his own main outcome among these 3 criteria.

DETAILED DESCRIPTION:
Raynaud's phenomenon (RP) is a clinical condition that follows an exaggerated vasoconstriction of extremities in response to a cold or emotional stress. Microvascular dysfunction and alteration of the endothelial NO-dependent vasodilatation pathway through NO synthases (NOS) represents one of the main mechanisms.

A pharmacological treatment in RP is proposed to patients when conservative measures are not efficient enough to control the symptoms: calcium channel blockers remains the first line, phosphodiesterase type 5 inhibitors as a second line treatment, while intravenous iloprost remains restricted to patients with digital ischaemia. Vasodilator therapies are commonly associated with side effects due to the non-specific systemic vasodilation that often result in permanent discontinuation. Many patients prefer complementary and alternative therapies, but none has proven its efficacy. Therefore, there is still room for improvement in the treatment of RP, and research is needed in this area.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18
* Active Raynaud's Phenomenon characterized by a clinical history of Raynaud's

  1. Primary RP or secondary to limited (LSSc), limited or diffuse cutaneous scleroderma (lcSSc or dcSSc) according to the criteria of Leroy and Medsger.
  2. At least 1 RP attacks per week and a specific finger patient picture in RP attack (assessed over the 2 weeks preceding inclusion)
* Stable disease over the previous two months (i.e. recent diagnosis of SSc will be excluded)
* Patients insured by a social security scheme or beneficiaries of such a scheme
* Patients who have dated and signed the informed consent form

Exclusion Criteria:

* Uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled angina
* Haemodynamic instability
* Pregnancy (or considering pregnancy in next 4 months) or breast feeding
* Subject in an exclusion period from another study,
* Subject under administrative or judicial supervision
* Subject not able to be contacted in case of emergency

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Raynaud Condition Score | first winter: inclusion visit week 2, week 7, week 13, week 19; second winter: inclusion visit week 2,week 7, week 13, week 19
  Change from baseline in the Raynaud's Condition score (RCS). RCS is participant's rating of difficulty considering number of attacks, duration, amount of pain, numbness, or other symptoms caused in the fingers (including painful sores) due to the Raynaud's phenomenon every day and impact of Raynaud's alone on use of hands every day. An 11 point Likert scale is used to rate the difficulty caused by the condition each day with 0 = no difficulty and 10 = extreme difficulty.
Frequency of RP | 7 days (An attack is defined as an episode of pallor or cyanosis (with or without pain,tingling or numbness). The number of attacks is self-reported every day and averaged over 7-day periods)
  number of RP attacks during treatment, as compared to placebo
Change in cumulative attack duration | first winter: inclusion visit week 2, week 7, week 13, week 19; second winter: inclusion visit week 2,week 7, week 13, week 19
  Mean duration of Raynaud's attacks for a time period was calculated as sum of recorded durations of attacks in the time period divided by total number of attacks in the time period where duration was recorded.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | first winter: week 2, 4, 5, 7, 13, 19; second winter: week 2, 4, 5, 7, 13, 19
  Mean duration of Raynaud's attacks for a time period was calculated as sum of recorded durations of attacks in the time period divided by total number of attacks in the time period where duration was recorded.
  It will be assessed through adverse events collected in the daily dairies cards.
Plasma concentration of L-arginine/ADMA ratio | first winter: week 2, 4, 5, 7; second winter: week 2, 4, 5, 7
  It will be quantified and compared under the 4 conditions.
Plasma concentration of nitrites | first winter: week 2, 4, 5, 7; second winter: week 2, 4, 5, 7
  It will be quantified and compared under the 4 conditions.
Plasma concentration of L-arginine | first winter: week 2, 4, 5, 7; second winter: week 2, 4, 5, 7
  It will be quantified and compared under the 4 conditions.
Urinary GMPc | first winter: week 2, 4, 5, 7; second winter: week 2, 4, 5, 7
  It will be quantified and compared under the 4 conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Cracowski, MD, Principal Investigator — Grenoble University Hospital, Clinical Pharmacology Department
Locations (1):
- Grenoble University Hospital, Grenoble, France